CLINICAL TRIAL: NCT00861744
Title: A Phase II, Randomized, Observer Blind, Controlled, Multicenter Study to Assess Immunogenicity and Antibody Persistence Following Vaccination With GSK's Candidate Combined Measles, Mumps, and Rubella Vaccine (MMR) Versus M-M-R® II as a First Dose, Both Administered Subcutaneously at 12-15 Months of Age, Concomitantly With Hepatitis A Vaccine (HAV), Varicella Vaccine (VV) and Pneumococcal Conjugate Vaccine (PCV) But at Separate Sites.
Brief Title: Immunogenicity of GSKs' MMR Vaccine (209762) vs. M-M-R® II, When Given With Routine Vaccines at 12-15 Months of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 111870; 2011-005860-31 (EudraCT Number)
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Results first posted 2011-11-04 (Estimated); Last update posted 2020-01-03 (Actual); Status verified 2019-12

CONDITIONS: Rubella; Mumps; Measles; Measles-Mumps-Rubella Vaccine
Keywords: Measles, Mumps, Rubella, Varicella Vaccine; Children; Immunogenicity; Safety; Humans; Combined Vaccine; Vaccines
MeSH Terms: conditions — Rubella; Mumps; Measles | interventions — Chickenpox Vaccine; Hepatitis A Vaccines; Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (4):
- Priorix 1 Group (Experimental): Subjects between 12 and 15 months of age at the time of study vaccination who received one dose of Priorix investigational vaccine (Lot 1) subcutaneously in the right upper arm. Subjects concomitantly received one dose of Havrix and Prevnar vaccines intramuscularly in the left and the right thigh, respectively and one dose of Varivax vaccine subcutaneously in the left upper arm. Subjects had previously received three doses of Prevnar vaccine within the first year of life with the third dose administered at least 30 days prior to enrollment and vaccination with study vaccines.
  Interventions: Biological: GSK Biological's investigational vaccine 209762; Biological: Varivax®; Biological: Havrix®; Biological: Prevnar®
- Priorix 2 Group (Experimental): Subjects between 12 and 15 months of age at the time of study vaccination who received one dose of Priorix investigational vaccine (Lot 2) subcutaneously in the right upper arm. Subjects concomitantly received one dose of Havrix and Prevnar vaccines intramuscularly in the left and the right thigh, respectively and one dose of Varivax vaccine subcutaneously in the left upper arm. Subjects had previously received three doses of Prevnar vaccine within the first year of life with the third dose administered at least 30 days prior to enrollment and vaccination with study vaccines.
  Interventions: Biological: GSK Biological's investigational vaccine 209762; Biological: Varivax®; Biological: Havrix®; Biological: Prevnar®
- Priorix 3 Group (Experimental): Subjects between 12 and 15 months of age at the time of study vaccination who received one dose of Priorix investigational vaccine (Lot 3) subcutaneously in the right upper arm. Subjects concomitantly received one dose of Havrix and Prevnar vaccines intramuscularly in the left and the right thigh, respectively and one dose of Varivax vaccine subcutaneously in the left upper arm. Subjects had previously received three doses of Prevnar vaccine within the first year of life with the third dose administered at least 30 days prior to enrollment and vaccination with study vaccines.
  Interventions: Biological: GSK Biological's investigational vaccine 209762; Biological: Varivax®; Biological: Havrix®; Biological: Prevnar®
- MMR-II Group (Active Comparator): Subjects between 12 and 15 months of age at the time of study vaccination who randomly received one dose of one of three different commercially-available lot of M-M-R II (Merck and Co.) vaccine subcutaneously in the right upper arm. Subjects concomitantly received one dose of Havrix and Prevnar vaccines intramuscularly in the left and the right thigh, respectively and one dose of Varivax vaccine subcutaneously in the left upper arm. Subjects had previously received three doses of Prevnar vaccine within the first year of life with the third dose administered at least 30 days prior to enrollment and vaccination with study vaccines.
  Interventions: Biological: M-M-R® II (Merck and Co); Biological: Varivax®; Biological: Havrix®; Biological: Prevnar®

INTERVENTIONS:
Biological: GSK Biological's investigational vaccine 209762 — Subcutaneous injection, one dose
  Arms: Priorix 1 Group; Priorix 2 Group; Priorix 3 Group
Biological: M-M-R® II (Merck and Co) — Subcutaneous injection, one dose
  Arms: MMR-II Group
Biological: Varivax® — Subcutaneous injection, one dose
Biological: Havrix® — Intramuscular injection, one dose
Biological: Prevnar® — Intramuscular injection, one dose

SUMMARY:
The purpose of this study is to compare two measles, mumps and rubella conjugate vaccines (manufactured by GSK and Merck and Company ) in terms of the immune response elicited and safety with a six month follow-up after first vaccination. Additionally, antibody persistence will be assessed one and two years after administration of MMR vaccine.

The Protocol Posting has been updated following Protocol amendment 1 and 2, Oct 2009.

ELIGIBILITY:
Inclusion Criteria:

* Subjects for whom the investigator believes their parents/guardians can and will comply with the requirements of the protocol (e.g. completion of the diary cards, return for follow-up visits) should be enrolled in the study.
* Male or female between 12 and 15 months of age (e.g. from age 12 months until the day before age 16 months) at the time of vaccination.
* Written informed consent obtained from the parent/guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Have previously received three doses of 7-valent pneumococcal conjugate vaccine within the first year of life with the third dose administered at least 30 days prior to enrolment and vaccination with study vaccines.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product (pharmaceutical product or device).
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol from 30 days prior to vaccination until 42 days after vaccination, except for influenza vaccine and Hib vaccine.
* Previous vaccination against measles, mumps, rubella and/or varicella.
* Previous vaccination against hepatitis A or receipt of a fourth dose of pneumococcal conjugate vaccine.
* History of measles, mumps, rubella, varicella/zoster and hepatitis A diseases.
* Known exposure to measles, mumps, rubella and/or varicella/zoster within 30 days prior to the start of the study.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination (no laboratory testing required), including human immunodeficiency virus (HIV) infection.
* A family history of congenital or hereditary immunodeficiency.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* Hypersensitivity to latex
* Major congenital defects or serious chronic illness.
* History of any neurologic disorders or seizures, including febrile seizures.
* Acute disease at the time of enrolment.
* Administration of polyclonal immunoglobulins and/or any blood products during the six months before entering the study or planned administration during the study period.

Ages: 12 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1259 (Actual)
Dates: Start 2009-06-03 (Actual); Primary Completion 2010-07-21 (Actual); Study Completion 2012-06-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (48):
- United States (45):
  - GSK Investigational Site, Tuscaloosa, Alabama
  - GSK Investigational Site, Conway, Arkansas
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Anaheim, California
  - GSK Investigational Site, Downey, California
  - GSK Investigational Site, Fresno, California
  - GSK Investigational Site, Huntington Beach, California
  - GSK Investigational Site, Paramount, California
  - GSK Investigational Site, Santa Ana, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Dalton, Georgia
  - GSK Investigational Site, Marietta, Georgia
  - GSK Investigational Site, Nampa, Idaho
  - GSK Investigational Site, DeKalb, Illinois
  - GSK Investigational Site, Arkansas City, Kansas
  - GSK Investigational Site, Bardstown, Kentucky
  - GSK Investigational Site, Bossier City, Louisiana
  - GSK Investigational Site, Metairie, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Kansas City, Missouri
  - GSK Investigational Site, Great Falls, Montana
  - GSK Investigational Site, Henderson, Nevada
  - GSK Investigational Site, Utica, New York
  - GSK Investigational Site, Cary, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Tulsa, Oklahoma
  - GSK Investigational Site, Gresham, Oregon
  - GSK Investigational Site, East Norriton, Pennsylvania
  - GSK Investigational Site, Rydal, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Bristol, Tennessee
  - GSK Investigational Site, Kingsport, Tennessee
  - GSK Investigational Site, Corpus Christi, Texas
  - GSK Investigational Site, Layton, Utah
  - GSK Investigational Site, Provo, Utah
  - GSK Investigational Site, Springville, Utah
  - GSK Investigational Site, St. George, Utah
  - GSK Investigational Site, West Jordan, Utah
  - GSK Investigational Site, Virginia Beach, Virginia
  - GSK Investigational Site, Huntington, West Virginia
- Puerto Rico (3):
  - GSK Investigational Site, Bayamón
  - GSK Investigational Site, San Germán
  - GSK Investigational Site, San Juan

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=3669

REFERENCES:
- [Background] Mufson MA, Diaz C, Leonardi M, Harrison CJ, Grogg S, Carbayo A, Carlo-Torres S, JeanFreau R, Quintero-Del-Rio A, Bautista G, Povey M, Da Costa C, Nicholson O, Innis BL. Safety and Immunogenicity of Human Serum Albumin-Free MMR Vaccine in US Children Aged 12-15 Months. J Pediatric Infect Dis Soc. 2015 Dec;4(4):339-48. doi: 10.1093/jpids/piu081. Epub 2014 Aug 7. PMID 26582873
- [Derived] Berry AA, Abu-Elyazeed R, Diaz-Perez C, Mufson MA, Harrison CJ, Leonardi M, Twiggs JD, Peltier C, Grogg S, Carbayo A, Shapiro S, Povey M, Baccarini C, Innis BL, Henry O. Two-year antibody persistence in children vaccinated at 12-15 months with a measles-mumps-rubella virus vaccine without human serum albumin. Hum Vaccin Immunother. 2017 Jul 3;13(7):1516-1522. doi: 10.1080/21645515.2017.1309486. Epub 2017 May 8. PMID 28481690
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111870 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was divided in 3 phases: the active phase (up to Day 42), the extended safety follow-up (ESFU) phase (up to Day 180) and the antibody persistence phase (up to Day 730).
Pre-assignment Details: The number of subjects enrolled was 1259. 39 subjects were enrolled in the study but did not receive a subject number and were never vaccinated.
Period: Overall Study
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Started | 304 | 304 | 304 | 308
Completed | 287 | 275 | 280 | 275
Not Completed | 17 | 29 | 24 | 33
Not completed — Adverse Event | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 7 | 19 | 17 | 12
Not completed — Withdrawal by Subject | 10 | 6 | 6 | 19
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Migration from study area | 0 | 3 | 1 | 0
Not completed — Blood draws | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group | Total
Number analyzed (Participants) | 304 | 304 | 304 | 308 | 1220
Age, Continuous [Mean (Standard Deviation); unit: Months] | 12.4 (0.75) | 12.4 (0.73) | 12.2 (0.56) | 12.4 (0.75) | 12.4 (0.70)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 156 | 144 | 157 | 139 | 596
  Male | 148 | 160 | 147 | 169 | 624

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Cut-off-value.
Description: Anti-measles virus antibody cut-off-value assessed was ≥ 200 milli-International Units per milliliter (mIU/mL). The analysis was performed on seronegative subjects. Seronegative subjects are subjects with anti-measles virus antibody concentrations <150 mIU/mL prior to vaccination.
Time Frame: At Day 42 after administration of a dose of Priorix vaccine.
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity, which included eligible subjects with pre- and post-vaccination serology results available.
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 247 | 240 | 240 | 249
Subjects | 245 | 236 | 236 | 248

2. Primary Outcome: Number of Subjects With Anti-mumps Virus Antibody Titer Equal to or Above the Cut-off-value.
Description: Anti-mumps virus antibody cut-off-value assessed was ≥ 51 Estimated Dose 50 (ED50). The analysis was performed on seronegative subjects. Seronegative subjects are subjects with anti-measles virus antibody concentrations <24 ED50 prior to vaccination.
Time Frame: At Day 42 after administration of a dose of Priorix vaccine.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 193 | 202 | 195 | 192
Subjects | 175 | 183 | 175 | 175

3. Primary Outcome: Number of Subjects With Anti-rubella Virus Antibody Concentrations Equal to or Above the Cut-off-value.
Description: Anti-rubella virus antibody cut-off-value assessed was ≥ 10 International Units per milliliter (IU/mL).
Time Frame: At Day 42 after administration of a dose of Priorix vaccine.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 247 | 238 | 239 | 249
Subjects | 244 | 235 | 233 | 249

4. Secondary Outcome: Number of Subjects With Anti-varicella Antibody Concentration Equal to or Above the Cut-off-value.
Description: Anti-varicella virus antibody cut-off-value assessed was ≥ 75 milli-International Units per milliliter (mIU/mL).
Time Frame: At Day 42 after administration of a dose of Varivax vaccine.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 245 | 238 | 240 | 246
Subjects | 240 | 230 | 230 | 241

5. Secondary Outcome: Anti-measles Virus Antibody Concentrations
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMCs) in mIU/mL. The analysis was performed on seronegative subjects. Seronegative subjects are subjects with anti-measles virus antibody concentrations <150 mIU/mL prior to vaccination.
Time Frame: At Day 42 after administration of a dose of Priorix vaccine.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 247 | 240 | 240 | 249
mIU/mL | 2798.7 [2544.8 to 3077.9] | 2878.2 [2607.0 to 3177.7] | 2593.1 [2350.3 to 2861.1] | 2949.5 [2698.4 to 3224.0]

6. Secondary Outcome: Anti-mumps Virus Antibody Concentrations
Description: Antibody concentrations are expressed as Geometric Mean Titer (GMT). The analysis was performed on seronegative subjects. Seronegative subjects are subjects with antibody titer < 24 ED50 prior to vaccination.
Time Frame: At Day 42 after administration of a dose of Priorix vaccine.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 193 | 202 | 195 | 192
Titers | 242.0 [204.5 to 286.5] | 265.0 [221.8 to 316.5] | 253.4 [213.4 to 300.9] | 267.6 [224.2 to 319.5]

7. Secondary Outcome: Anti-rubella Virus Antibody Concentrations
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMCs) in IU/mL. The analysis was performed on seronegative subjects. Seronegative subjects are subjects with anti-rubella virus antibody concentrations <4 IU/mL prior to vaccination.
Time Frame: At Day 42 after administration of a dose of Priorix vaccine.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 247 | 238 | 239 | 249
IU/mL | 72.2 [65.6 to 79.6] | 77.7 [70.4 to 85.7] | 68.2 [61.8 to 75.3] | 89.4 [81.4 to 98.2]

8. Secondary Outcome: Anti-S. Pneumoniae Antibody Concentrations (by Serotype).
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMCs) in µg/mL.
Time Frame: At Day 42 after vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 128 | 127 | 128 | 126
µg/mL
  Anti-S.PNEU-4 | 3.57 [3.04 to 4.20] | 3.72 [3.21 to 4.31] | 3.40 [2.88 to 4.00] | 3.80 [3.17 to 4.56]
  Anti-S. PNEU-6B | 5.68 [4.78 to 6.76] | 5.87 [5.02 to 6.87] | 5.41 [4.66 to 6.28] | 7.22 [6.28 to 8.29]
  Anti-S.PNEU 9V | 6.56 [5.66 to 7.60] | 7.30 [6.35 to 8.38] | 5.81 [4.97 to 6.78] | 7.80 [6.81 to 8.93]
  Anti-S.PNEU-14 | 9.23 [8.03 to 10.61] | 8.33 [7.30 to 9.51] | 7.58 [6.55 to 8.76] | 7.97 [6.95 to 9.14]
  Anti-S.PNEU-18 C | 6.20 [5.30 to 7.26] | 6.62 [5.76 to 7.60] | 6.15 [5.25 to 7.21] | 6.73 [5.74 to 7.91]
  Anti-S.PNEU-19 F | 2.42 [2.05 to 2.85] | 2.46 [2.11 to 2.88] | 2.34 [2.00 to 2.73] | 2.59 [2.23 to 3.00]
  Anti-S.PNEU-23 F | 9.34 [7.76 to 11.25] | 9.27 [7.82 to 10.99] | 8.33 [6.88 to 10.10] | 11.49 [9.67 to 13.66]

9. Secondary Outcome: Anti-varicella Antibody Concentrations.
Description: Antibody concentrations are expressed as Geometric Mean Titers (GMT). The analysis was performed on seronegative subjects. Seronegative subjects are subjects with antibody concentration < 25 mIU/mL prior to vaccination.
Time Frame: At Day 42 after administration of a dose of Varivax vaccine.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 245 | 238 | 240 | 246
mIU/mL | 245.5 [229.0 to 263.3] | 235.2 [217.4 to 254.4] | 236.0 [218.0 to 255.5] | 255.9 [240.4 to 272.4]

10. Secondary Outcome: Anti-hepatitis A Virus Antibody Concentrations.
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMCs) in mIU/mL. The analysis was performed on seronegative subjects. Seronegative subjects are subjects with anti-hepatitis A virus antibody concentrations <15 mIU/mL prior to vaccination.
Time Frame: At Day 42 after administration of a dose of Havrix vaccine.
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 117 | 112 | 111 | 124
mIU/mL | 33.8 [28.8 to 39.6] | 39.2 [33.1 to 46.5] | 39.4 [32.7 to 47.5] | 42.1 [35.8 to 49.6]

11. Secondary Outcome: Number of Subjects With Anti-hepatitis A Antibody Concentrations Equal to or Above the Cut-off-value.
Description: Anti-hepatitis A antibody cut-off-value assessed was ≥15 milli-International Units per milliliter (mIU/mL).
Time Frame: At Day 42 after administration of a dose of Havrix vaccine.
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 117 | 112 | 111 | 124
Subjects | 98 | 99 | 94 | 110

12. Secondary Outcome: Anti-S. Pneumoniae Antibody Concentrations (by Serotype).
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMCs) in µg/mL.
Time Frame: At Day 0 before vaccination
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: µg/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 129 | 130 | 130 | 119
µg/mL
  Anti-S.PNEU-4 | 0.54 [0.46 to 0.65] | 0.61 [0.52 to 0.72] | 0.67 [0.58 to 0.78] | 0.67 [0.56 to 0.81]
  Anti-S.PNEU-6B | 0.53 [0.43 to 0.66] | 0.57 [0.46 to 0.70] | 0.52 [0.43 to 0.64] | 0.67 [0.56 to 0.80]
  Anti-S.PNEU-9V | 1.01 [0.85 to 1.20] | 1.13 [0.97 to 1.32] | 1.04 [0.88 to 1.23] | 1.26 [1.06 to 1.49]
  Anti-S.PNEU-14 | 3.01 [2.60 to 3.47] | 2.82 [2.42 to 3.28] | 2.54 [2.21 to 2.92] | 2.76 [2.38 to 3.20]
  Anti-S.PNEU-18C | 0.88 [0.74 to 1.03] | 0.97 [0.83 to 1.13] | 0.97 [0.83 to 1.14] | 1.00 [0.86 to 1.15]
  Anti-S.PNEU-19F | 0.40 [0.32 to 0.50] | 0.40 [0.33 to 0.50] | 0.44 [0.36 to 0.53] | 0.45 [0.37 to 0.56]
  Anti-S.PNEU-23 F | 0.64 [0.51 to 0.82] | 0.63 [0.51 to 0.77] | 0.65 [0.52 to 0.81] | 0.85 [0.67 to 1.08]

13. Secondary Outcome: Number of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Anti-measles virus antibody cut-off-value assessed was ≥ 200 milli-International Units per milliliter (mIU/mL).
Time Frame: At 1 year post-vaccination
Population: The analysis was based on the according-to-protocol (ATP) cohort for persistence at Year 1, which included all eligible subjects who received study vaccine/comparator, for whom data concerning immunogenicity outcome measures were available At Day 0, Day 42 post-vaccination, and Year 1 post-vaccination and who complied with blood sampling schedules.
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 213 | 215 | 218 | 210
Subjects | 211 | 211 | 218 | 209

14. Secondary Outcome: Number of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Cut-off-value
Description: Anti-measles virus antibody cut-off-value assessed was ≥ 200 milli-International Units per milliliter (mIU/mL).
Time Frame: At 2 years post-vaccination
Population: The analysis was based on the according-to-protocol (ATP) cohort for persistence at Year 2, which included all eligible subjects who received study vaccine/comparator, for whom data concerning immunogenicity outcome measures were available At Day 0, Day 42 post-vaccination, and Year 2 post-vaccination and who complied with blood sampling schedules.
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 171 | 159 | 169 | 166
Subjects | 171 | 159 | 168 | 166

15. Secondary Outcome: Anti-measles Virus Antibody Concentrations
Description: as for outcome 5
Time Frame: At 2 years post-vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 171 | 159 | 169 | 166
mIU/mL | 3361.1 [2922.3 to 3865.6] | 3963.8 [3479.3 to 4515.7] | 3360.3 [2923.3 to 3862.7] | 4022.1 [3507.7 to 4611.9]

16. Secondary Outcome: Anti-measles Virus Antibody Concentrations
Description: Antibody concentrations were expressed as Geometric Mean Concentrations (GMCs) in mIU/mL. The analysis was performed on seronegative subjects. Seronegative subjects are subjects with anti-measles virus antibody concentrations <150 mIU/mL prior to vaccination.
Time Frame: At 1 year post-vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 213 | 215 | 218 | 210
mIU/mL | 3224.3 [2840.1 to 3660.5] | 3708.2 [3226.2 to 4262.2] | 3534.7 [3139.9 to 3979.1] | 3828.1 [3371.3 to 4346.7]

17. Secondary Outcome: Number of Subjects Reporting Investigator-confirmed Measles/Rubella-like Rash and Varicella-like Rash.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: The analysis of safety was performed on the Total Vaccinated cohort, which included all subjects with the vaccine administration documented and symptom sheet completed, only on subjects that reported the specific symptom.
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 283 | 275 | 283 | 277
Subjects
  Varicella like | 0 | 4 | 0 | 0
  Measles/Rubella like | 6 | 7 | 5 | 5

18. Secondary Outcome: Number of Subjects Reporting Febrile Convulsions
Description: Timing of febrile convulsions: events occured on Day 29 in the Priorix 2 Group and Day 0 in the MMR II Group. All cases of febrile convulsions were case of meningism.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 17
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 283 | 275 | 283 | 277
Subjects | 0 | 1 | 0 | 1

19. Secondary Outcome: Anti-mumps Virus Antibody Titers (Enhanced Plaque Reduction Neutralization (PRN))
Description: Antibody titers were expressed as Geometric Mean Titer (GMT). The analysis was performed on seronegative subjects. Seronegative subjects are subjects with antibody titer < 24 ED50 prior to vaccination.
Time Frame: At 1 year post-vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 189 | 186 | 189 | 183
Titers | 162.8 [141.8 to 186.9] | 188.3 [162.4 to 218.3] | 176.2 [152.6 to 203.3] | 185.5 [163.5 to 210.6]

20. Secondary Outcome: Number of Subjects Reporting Other Rash.
Description: Other rash = not confirmed by the investigator to be either measles/rubella-like or varicella-like in nature
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 17
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 283 | 275 | 283 | 277
Subjects
  Localized or generalized | 72 | 74 | 60 | 60
  With fever | 26 | 29 | 23 | 23
  Grade 3 | 11 | 10 | 6 | 6
  Related | 9 | 14 | 6 | 6

21. Secondary Outcome: Number of Subjects With Anti-mumps Virus Antibody Titers Above the Cut-off Value (Enhanced PRN)
Description: Anti-mumps virus antibody cut-off-value assessed was ≥ 51 ED50.
Time Frame: At 1 year post-vaccination
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 189 | 186 | 189 | 183
Subjects | 169 | 170 | 171 | 170

22. Secondary Outcome: Number of Subjects With Anti-rubella Virus Antibody Concentrations Equal to or Above the Cut-off-value.
Description: Anti-rubella virus antibody cut-off-value assessed was ≥ 10 International Units per milliliter (IU/mL). The analysis was performed on seronegative subjects. Seronegative subjects are subjects with anti-rubella virus antibody concentrations <4 IU/mL prior to vaccination.
Time Frame: At 1 year post-vaccination
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 213 | 214 | 218 | 210
Subjects | 212 | 213 | 217 | 210

23. Secondary Outcome: Number of Subjects With Anti-rubella Virus Antibody Concentrations Equal to or Above the Cut-off-value.
Description: Anti-rubella virus antibody cut-off-value assessed was ≥ 10 International Units per milliliter (IU/mL).
Time Frame: At 2 years post-vaccination
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 171 | 158 | 168 | 166
Subjects | 171 | 158 | 168 | 166

24. Secondary Outcome: Anti-rubella Virus Antibody Concentrations
Description: as for outcome 7
Time Frame: At 1 year post-vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 213 | 214 | 218 | 210
IU/mL | 138.1 [125.3 to 152.2] | 145.4 [132.0 to 160.1] | 136.5 [123.5 to 150.9] | 166.8 [151.5 to 183.6]

25. Secondary Outcome: Anti-rubella Virus Antibody Concentrations
Description: as for outcome 7
Time Frame: At 2 years post-vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 171 | 158 | 168 | 166
IU/mL | 78.0 [69.7 to 87.2] | 79.5 [71.7 to 88.2] | 81.7 [73.8 to 90.4] | 93.1 [83.6 to 103.6]

26. Secondary Outcome: Number of Subjects Reporting Fever.
Description: fever is assessed for temperature ≥38°C/100.4°F and >39.5°C/103.1°F as measured rectally.
Time Frame: During the 15-day (Days 0-14) and 43 days (Days 0-42) post-vaccination period
Population: as for outcome 17
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 283 | 275 | 283 | 277
Subjects
  Day 15 (N= 283; 275; 283; 277) ≥38.0°C | 65 | 79 | 64 | 56
  Day 15 (N= 283; 275; 283; 277) >39.5°C | 10 | 7 | 9 | 8
  Day 43 (N= 283; 275; 283; 277) ≥38.0°C | 103 | 104 | 104 | 85
  Day 43 (N= 283; 275; 283; 277) >39.5°C | 20 | 14 | 18 | 13

27. Secondary Outcome: Number of Subjects With Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: as for outcome 17
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 282 | 274 | 282 | 274
Subjects
  Pain | 70 | 70 | 79 | 67
  Redness | 45 | 47 | 41 | 47
  Swelling | 20 | 26 | 19 | 15

28. Secondary Outcome: Number of Subjects Reporting Medically Attended Visit (MAEs)
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: The analysis of safety was performed on the Total Vaccinated cohort, which included all subjects with the vaccine administration documented.
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 304 | 304 | 304 | 308
Subjects | 99 | 99 | 97 | 107

29. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs).
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any = the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 304 | 304 | 304 | 308
Subjects | 170 | 153 | 164 | 169

30. Secondary Outcome: Number of Subjects Reporting Investigator-confirmed Parotid/Salivary Gland Swelling.
Description: Swelling with accompanying general symptoms
Time Frame: During the 43-day (Days 0-42) post-vaccination period
Population: as for outcome 17
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 283 | 275 | 283 | 277
Subjects | 3 | 3 | 5 | 2

31. Secondary Outcome: Number of Subjects With Solicited General Symptoms.
Description: Assessed solicited general symptoms were drowsiness, irritability and loss of appetite. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During the 15-day (Days 0-14) post-vaccination period
Population: as for outcome 17
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 283 | 275 | 283 | 277
Subjects
  Any drowsiness | 133 | 106 | 113 | 109
  Any irritability | 180 | 141 | 150 | 153
  Any loss of appetite | 111 | 77 | 110 | 94

32. Secondary Outcome: Number of Subjects Reporting New Onset Chronic Illnesses (NOCIs).
Description: NOCIs included autoimmune disorders, asthma, type I diabetes, allergies.
Time Frame: From Day 0 to Day 180 after vaccination
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 304 | 304 | 304 | 308
Subjects | 5 | 2 | 4 | 2

33. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to Day 180 after vaccination
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 304 | 304 | 304 | 308
Subjects | 1 | 6 | 7 | 9

34. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs).
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 180 to Day 730 after vaccination
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 304 | 304 | 304 | 308
Subjects | 0 | 0 | 0 | 1

35. Secondary Outcome: Number of Subjects Reporting Conditions Prompting Emergency Room (ER) Visits.
Time Frame: From Day 0 to Day 180 after vaccination
Population: as for outcome 28
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 304 | 304 | 304 | 308
Subjects | 27 | 28 | 22 | 26

36. Secondary Outcome: Anti-mumps Virus Antibody Titers (Unenhanced PRN)
Description: Antibody titers were expressed as Geometric Mean Titer (GMT).
Time Frame: At 1 year post-vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 196 | 205 | 211 | 195
Titer | 31.0 [24.1 to 39.9] | 46.1 [36.2 to 58.7] | 39.3 [31.0 to 50.0] | 46.6 [36.6 to 59.3]

37. Secondary Outcome: Number of Subjects With Anti-mumps Virus Antibody Titers Above the Cut-off Value (Unenhanced PRN)
Description: Anti-mumps virus antibody cut-off-value assessed was ≥ 4 Estimated Dose 50 (ED50).
Time Frame: At 1 year post-vaccination
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 196 | 205 | 211 | 195
Subjects | 173 | 186 | 184 | 173

38. Secondary Outcome: Anti-mumps Virus Antibody Titers (Unenhanced PRN)
Description: Antibody concentrations are expressed as Geometric Mean Titer (GMT).
Time Frame: At 2 years post-vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 157 | 144 | 157 | 152
Titer | 43.4 [33.4 to 56.3] | 48.9 [37.7 to 63.5] | 57.4 [45.7 to 72.2] | 60.7 [47.6 to 77.5]

39. Secondary Outcome: Number of Subjects With Anti-mumps Virus Antibody Titers Above the Cut-off Value (Unenhanced PRN)
Description: Anti-mumps virus antibody cut-off-value assessed was ≥ 4 Estimated Dose 50 (ED50).
Time Frame: At 2 years post-vaccination
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 157 | 144 | 157 | 152
Subjects | 144 | 134 | 152 | 144

40. Secondary Outcome: Anti-mumps Virus Antibody Concentrations (Pharmaceutical Product Development (PPD) ELISA)
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMC) in ELISA units per milliliter (EU/mL). The analysis was performed on seronegative subjects. Seronegative subjects are subjects with anti-rubella virus antibody concentrations <5 EU/mL prior to vaccination.
Time Frame: At 1 year post-vaccination
Population: as for outcome 13
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 170 | 173 | 179 | 170
EU/mL | 47.3 [39.2 to 57.1] | 42.9 [36.4 to 50.6] | 42.5 [35.9 to 50.3] | 58.6 [50.6 to 67.8]

41. Secondary Outcome: Number of Subjects With Anti-mumps Virus Antibody Concentrations Above the Cut-off Value (PPD ELISA)
Description: Anti-mumps virus antibody cut-off-value assessed was ≥ 10 ELISA units per milliliter (EU/mL)
Time Frame: At 1 year post-vaccination
Population: as for outcome 13
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 170 | 173 | 179 | 170
Subjects | 155 | 159 | 162 | 164

42. Secondary Outcome: Anti-mumps Virus Antibody Concentrations (PPD ELISA)
Description: as for outcome 40
Time Frame: At 2 years post-vaccination
Population: as for outcome 14
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 136 | 130 | 141 | 140
EU/mL | 47.8 [40.2 to 56.9] | 50.2 [42.1 to 59.9] | 54.0 [46.1 to 63.3] | 59.2 [50.1 to 70.0]

43. Secondary Outcome: Number of Subjects With Anti-mumps Virus Antibody Concentrations Above the Cut-off Value (PPD ELISA)
Description: Anti-mumps virus antibody cut-off-value assessed was ≥ 10 ELISA units per milliliter (EU/mL)
Time Frame: At 2 years post-vaccination
Population: as for outcome 14
Measure: Number; unit: Subjects
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
Number analyzed (Participants) | 136 | 130 | 141 | 140
Subjects | 128 | 125 | 136 | 134

ADVERSE EVENTS:
Time Frame: Solicited symptoms: During the 4-day (Days 0-3) post-vaccination period. Unsolicited AEs: During the 43-day (Days 0-42) post vaccination period. SAEs: the entire study period (Day 0-Day 730).
Description: Solicited symptoms were only assessed on subjects returning the symptom sheet.
Arm/Group | Priorix 1 Group | Priorix 2 Group | Priorix 3 Group | MMR-II Group
All-Cause Mortality (participants affected / at risk) | 0/304 | 0/304 | 0/304 | 0/308
Serious Adverse Events (participants affected / at risk) | 1/304 | 7/304 | 8/304 | 10/308
Other Adverse Events (participants affected / at risk) | 240/304 | 216/304 | 219/304 | 221/308
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Priorix 1 Group (N=304) | Priorix 2 Group (N=304) | Priorix 3 Group (N=304) | MMR-II Group (N=308)
Bronchiolitis (Infections and infestations) | 1 | 1 | 0 | 2 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Hypoxia (General disorders) | 0 | 0 | 0 | 2 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 1 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Croup infectious (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Inflenza like illness (General disorders) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Otitis media acute (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Pyrexia (General disorders) | 0 | 0 | 1 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Rash (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Respiratory syncitial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Ataxia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — Numbers correspond to all available data at the time of analysis of the active phase of the study.
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — From the beginning of the study (Day 0) up to Day 180.
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 — From the beginning of the study (Day 0) up to Day 180.
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 — From the beginning of the study (Day 0) up to Day 180.
Intussusception (Gastrointestinal disorders) | 0 | 0 | 1 | 0 — From the beginning of the study (Day 0) up to Day 180.
Influenza like illness (General disorders) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Pyrexia (General disorders) | 0 | 0 | 1 | 0 — From the beginning of the study (Day 0) up to Day 180.
Bronchiolitis (Infections and infestations) | 1 | 1 | 0 | 2 — From the beginning of the study (Day 0) up to Day 180.
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 1 — From the beginning of the study (Day 0) up to Day 180.
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 — From the beginning of the study (Day 0) up to Day 180.
Coxsackie viral infection (Infections and infestations) | 0 | 0 | 1 | 0 — From the beginning of the study (Day 0) up to Day 180.
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 1 | 0 — From the beginning of the study (Day 0) up to Day 180.
H1N1 influenza (Infections and infestations) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 — From the beginning of the study (Day 0) up to Day 180.
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Staphylococcal infection (Infections and infestations) | 0 | 1 | 0 | 0 — From the beginning of the study (Day 0) up to Day 180.
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Ataxia (Nervous system disorders) | 0 | 1 | 0 | 0 — From the beginning of the study (Day 0) up to Day 180.
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 — From the beginning of the study (Day 0) up to Day 180.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 — From the beginning of the study (Day 0) up to Day 180.
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 — From the beginning of the study (Day 0) up to Day 180.
Extremity necrosis (Vascular disorders) | 0 | 1 | 0 | 0 — From the beginning of the study (Day 0) up to Day 180.
Nephroblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 — SAE reported between Day 180 and Day 730 post-vaccination.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Priorix 1 Group (N=304) | Priorix 2 Group (N=304) | Priorix 3 Group (N=304) | MMR-II Group (N=308)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Acarodermatitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Acute tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aggression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Aphthous stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Arthropod sting (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (2) | 0 (0)
Auricular pseudocyst (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacterial test negative (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Blood iron decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bowel movement irregularity (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 3 (3) | 4 (4)
Bronchiolitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 5 (5)
Bronchitis (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Bronchitis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Burns second degree (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Cardiac murmur (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Eye disorders) | 9 (9) | 3 (3) | 0 (0) | 4 (4)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1) | 4 (5) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 25 (28) | 21 (24) | 16 (17) | 19 (19)
Croup infectious (Infections and infestations) | 4 (5) | 3 (3) | 6 (6) | 3 (3)
Crying (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Dark circles under eyes (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 111 (112) | 77 (78) | 110 (111) | 95 (96)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 25 (29) | 24 (29) | 19 (21) | 21 (22)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Discomfort (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drooling (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 3 (3)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 3 (3) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 46 (46) | 48 (49) | 43 (43) | 49 (49)
Eustachian tube dysfunction (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye allergy (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Eye swelling (Eye disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Faeces discoloured (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 2 (3) | 1 (1) | 2 (3) | 2 (2)
Fungal infection (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 5 (5) | 2 (2) | 5 (5)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Genital cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gynaecomastia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (3) | 2 (2) | 2 (5) | 5 (5)
Herpangina (Infections and infestations) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperpyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2) | 1 (2) | 2 (2)
Impetigo (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infected bites (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 2 (2) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Injection site bruising (General disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Injection site induration (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site mass (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site swelling (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (3) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 181 (185) | 142 (142) | 150 (152) | 153 (154)
Ketonuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Laryngomalacia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lethargy (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Middle insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Milk allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Molluscum contagiosum (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Mouth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Multiple allergies (Immune system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 (8) | 13 (13) | 9 (9) | 10 (11)
Nasal disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (11) | 8 (9) | 13 (14) | 9 (9)
Oedema peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media (Infections and infestations) | 25 (25) | 25 (26) | 29 (31) | 24 (26)
Otitis media acute (Infections and infestations) | 9 (10) | 10 (13) | 8 (8) | 5 (5)
Otitis media chronic (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Pain (General disorders) | 72 (72) | 70 (70) | 79 (79) | 68 (69)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1)
Pallor (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Penile adhesion (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 12 (12) | 7 (7) | 10 (10) | 6 (6)
Pharyngitis streptococcal (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 3 (3)
Pneumonia (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Polydipsia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 7 (7) | 4 (5) | 6 (8) | 4 (4)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 22 (27) | 17 (22) | 21 (25) | 13 (13)
Seasonal allergy (Immune system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus operation (Surgical and medical procedures) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 3 (3) | 5 (5) | 4 (5) | 3 (3)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 133 (133) | 106 (106) | 113 (114) | 109 (110)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Streptococcal infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling (General disorders) | 22 (22) | 26 (26) | 20 (20) | 15 (15)
Teething (Gastrointestinal disorders) | 35 (40) | 35 (41) | 37 (47) | 35 (40)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tongue disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Tooth discolouration (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (2) | 2 (7)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 40 (40) | 22 (25) | 39 (40) | 43 (46)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site bruise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 7 (7) | 8 (8) | 9 (9) | 11 (11)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral rash (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 13 (15) | 11 (13) | 13 (14) | 12 (13)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 4 (4) | 4 (4) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.